CLINICAL TRIAL: NCT06035861
Title: Investigating the Relationship Between Endothelial Cell Activation and Total Pulmonary Resistance in Pulmonary Artery Hypertension (PAH)
Brief Title: Endothelial Cell Activation and Total Pulmonary Resistance in PAH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22HH7807
Record Dates: First submitted 2023-08-30; First posted 2023-09-13 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Artery Hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension | interventions — N-benzyl-N-ethyl-2-(7,8-dihydro-7-methyl-8-oxo-2-phenyl-9H-purin-9-yl)acetamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XBD173 (Experimental): 6 weeks exposure to XBD173
  Interventions: Drug: XBD173

INTERVENTIONS:
Drug: XBD173 — Participants will be treated with XBD173 90mg twice daily for 6 weeks
  Other Names: AC5216

SUMMARY:
To determine whether changes in endothelial cell dysfunction are associated with changes in total pulmonary resistance in patients with pulmonary arterial hypertension

DETAILED DESCRIPTION:
Patients with PAH will be exposed to XBD173. Markers of endothelial cell dysfunction and activation will be measured in the plasma, and changes in total pulmonary resistance will be meausured with an implantable monitor

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 18-75 years old
2. PAH which is: idiopathic; PAH heritable; PAH associated with connective tissue disease; PAH after ≥ 1 year repair of congenital systemic to pulmonary shunt; or PAH associated with anorexignes or other drugs.
3. Resting mean pulmonary artery pressure ≥25 mmHg, pulmonary capillary wedge pressure ≤15 mmHg, PVR >5 wood units, and normal or reduced cardiac output, as measured by a previous right heart catheterisation (RHC).
4. Have an insertable FDA/CE cardiac rhythm monitor and pulmonary artery pressure monitor that captures cardiopulmonary haemodynamics and daily activity.
5. Six-minute walking distance >50m at entry
6. Stable on an unchanged PAH therapeutic regime comprising at least 2 therapies licensed for PAH (any combination of endothelin receptor antagonist, phosphodiesterase inhibitor or prostacyclin analogue) for at least 1 month prior to screening
7. Subjects willing to be genotyped for genes that influence XBD173 activity
8. Able to provide written informed consent prior to any study mandated procedures
9. Contraception: Fertile females (women of childbearing potential) are eligible to participate after a negative highly sensitive pregnancy test, if they are taking a highly effective method of contraception other than the oral contraceptive pill during treatment and until the end of relevant systemic exposure

Exclusion Criteria:

1. Unable to provide informed consent and/or are non-fluent speakers of the English language
2. Hypersensitivity to XBD173 or to any of the excipients
3. Clinically-significant renal disease (confirmed by creatinine clearance <30 ml/min per 1.73m2)
4. Clinically-significant liver disease (confirmed by serum transaminases >2 times than upper normal limit)
5. Anaemia confirmed by haemoglobin concentration <10 g/dl
6. Individuals known to have haemoglobinopathy sickle cell disease, thalassaemia
7. Hospital admission related to PAH or change in PAH therapy within 3 months prior to screening
8. History of left-sided heart disease and/or clinically significant cardiac disease, including but not limited to any of the following:

   1. Aortic or mitral valve disease (stenosis or regurgitation) defined as greater than mild aortic insufficiency, mild aortic stenosis, mild mitral stenosis, moderate mitral regurgitation
   2. Mechanical or bioprosthetic cardiac valve
   3. Pericardial constriction, effusion with tamponade physiology, or abnormal left atrial size.
   4. Restrictive or congestive cardiomyopathy
   5. Left ventricular ejection fraction ≤50% (measured in echocardiogram at screening)
   6. Symptomatic coronary disease
   7. Significant (2+ for regurgitation) valvular disease other than tricuspid or pulmonary regurgitation
   8. Acutely decompensated left heart failure within 1 month of screening
   9. History of untreated obstructive sleep apnoea
9. Evidence of significant lung disease on high-resolution CT (if available) or recent (performed within 12 months) lung function, where FEV1 < 50% predicted and FVC < 70% predicted, and DLCO (or TLCO) < 50% predicted if any CT abnormalities; judged by the Site Physician
10. Patients with a history of uncontrolled systemic hypertension
11. Acute infection (including eye, dental, and skin infections)
12. Chronic inflammatory disease including HIV, and Hepatitis B
13. Women of childbearing potential who are pregnant or breastfeeding (if applicable)
14. Patients who have received an Investigational Medicinal Product (IMP) within 5 half-lives of the last dose of the IMP or 1 month (which ever is greater) before the baseline visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Percentage change in plasma sVCAM1, e-selectin, GDF-15 and NT-proBNP | 6 weeks
  Percentage change in plasma markers
Percentage change in total pulmonary resistance | 6 weeks
  Percentage change in total pulmonary resistance

IPD SHARING:
Plan to Share IPD: No